CLINICAL TRIAL: NCT00399815
Title: Noninvasive Evaluation of Hepatic Fibrosis in Chronic Hepatitis C
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Prof Yves Horsmans, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Other Study IDs: ELASTO2
Record Dates: First submitted 2006-11-14; First posted 2006-11-15 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Hepatitis C, Chronic
Keywords: Chronic viral hepatitis C; HCV RNA; Fibroscan; Fibrotest; hepatic elastography by MRI
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — liver biopsy serum
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic viral hepatitis C is a frequent liver disease. It is associated with variable degree of hepatic fibrosis. To date, liver histology is still regarded as the gold standard to detect, diagnose and quantify liver fibrosis. This requires to perform a liver biopsy. Severe complications are associated to this procedure in 0.01 to 0.1% of cases. Because of this, the repetition of the biopsy to evaluate the progression of the disease or the response to treatment poses ethical questions. Also, liver biopsy only explore a minimal portion of the liver and liver fibrosis, which is not homogeneous, may be under- or over-estimated.

To avoid risks linked to invasive technique and sampling errors associated to liver biopsy, efforts are being made to develop non-invasive technology to detect and quantitate liver fibrosis.

In this study we will perform in patients with chronic hepatitis C, serum tests, fibroscan (elastography of liver parenchyma determined by ultra-sounds), and elastography of liver parenchyma by MRI.

This study will allow

* to determine whether non-invasive tests effectively measure liver fibrosis
* to compare each non-invase test with results of liver biopsy
* to determine whether a non-invasive test or a combination of non invasive tests may be used to accurately evaluate liver fibrosis in patients with chronic hepatitis C.

ELIGIBILITY:
Inclusion Criteria:

* alteration of liver function tests (ALT, AST)
* HCV RNA positive

Exclusion Criteria:

* clotting disorder
* ongoing treatment with anti-coagulant or anti-aggregant
* advanced or decompensated cirrhosis (Child-Pugh class C)
* hepatocellular carcinoma
* other cancer
* history of surgery for brain aneurysm
* pace maker or defibrillator
* ocular metal foreign body

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic hepatitis C
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2006-06; Primary Completion 2009-05 (Actual); Study Completion 2010-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yves J Horsmans, M.D., Ph.D., Study Director — Cliniques Universitaires StLuc, Université catholique de Louvain (UCL), Brussels, Belgium
Locations (1):
- Cliniques Universitaires StLuc, Université catholique de Louvain (UCL), Brussels, Belgium